CLINICAL TRIAL: NCT04516889
Title: Evaluating Safety and Efficacy of a Modified Technique of Scleral Fixation Intraocular Lens Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kam Ka Wai, Associate Consultant, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol V4.0
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Aphakia; Cataract
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention arm will undergo the modified sutured SFIOL technique with double Prolene sutures instead of a single Prolene suture
  Interventions: Procedure: Doubled sutured SFIOL

INTERVENTIONS:
Procedure: Doubled sutured SFIOL — Recruited subjects would undergo implantation of SFIOL with the modified technique under either local or general anesthesia. The surgeon would mark the sclerotomies as per routine sutured SFIOL at 2mm behind the nasal and temporal limbus, followed by passage of 2 pairs of prolene sutures. The intraocular lens with islets would be implanted into the posterior chamber and sutured to the sclera as per single suture SFIOL.

SUMMARY:
Cataract is the leading cause of blindness globally and cataract surgery with the implantation of intraocular lens (IOL) is the most commonly performed operation worldwide. After removal of the cataract, an IOL is usually implanted within the capsular bag. However, endocapsular implantation of IOL is not always feasible due to inadequate zonular or capsular support, intraoperative posterior capsule rupture, or in primary intracapsular cataract extraction. Predisposing factors including prior ocular trauma, intravitreal injection or intraocular surgery, co-existing ocular comorbidities like chronic uveitis, pseudoexfoliation syndrome, may increase the risk of failure of in-the-bag implantation.

In such situation, the surgeons may consider implanting the IOL in the anterior chamber, ciliary sulcus, or using fixation techniques. In Asian eyes, the anterior chambers are often shallow and placement in anterior chamber may accelerate corneal endothelial cell loss leading to corneal decompensation, or worsen pre-existing glaucoma. Placement in the ciliary sulcus depends on the amount and integrity of the capsular remnant, and inadequate support may result in dislocation of the IOL. In recent years, newer forms of scleral fixation of IOL using glue or glue-less approach, although these procedure appeared to be simpler, the long-term stability of these IOL have not been evaluated against conventional approach with suture fixation. The main limitations of suture fixation technique are related to the sutures either intraoperatively (e.g. entanglement, failure to rotate and bury the suture knot) or postoperatively (breakage, dissolution of suture with time), and the learning curve required for surgeons in training.

Our study aims to study the efficacy and safety of a modified technique of scleral fixation of an intraocular lens in the posterior chamber.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with phacodonesis, lens subluxation, insufficient capsular or zonular support, or surgical aphakia without adequate ciliary sulcus who are listed for scleral fixation intraocular lens implantation.

Exclusion Criteria:

* Patients with previous corneal transplantation surgery or undergoing concomitant corneal transplantation at the time of scleral fixation intraocular lens implantation.
* Patients undergoing concomitant vitreoretinal surgery at the time of intraocular lens implantation.
* Monocular patients, or patients whose fellow eye had vision of equal or less than 20/200.
* Patients who could not comprehend the risks and benefits of the surgery and/or the research study, including mentally incapacitated persons.
* Patients with pre-existing macular pathologies including macular oedema, haemorrhage, degeneration or scar.
* Patients with pre-existing iris abnormalities including aniridia, corectopia, extensive anterior synechiae formation resulting in inability to measure the IOL tilting postoperatively.
* Patients with significantly reduced corneal endothelial cell density (of < 1000 cells/mm2) preoperatively which may necessitate a corneal transplantation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of eyes with intraoperative, early (within 1 week) and late (at 12 months) postoperative complications following this modified technique of intraocular lens fixation. | up to 12 months
  Complication Rate

SECONDARY OUTCOMES:
Unaided and corrected visual acuities | up to 12 months
  Visual acuities
Intraocular lens tilting | up to 12 months
  Anterior segment optical coherence tomography
endothelial cell status | up to 12 months
  specular microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Alvin L Young, Principal Investigator — Prince of Wales Hospital

IPD SHARING:
Plan to Share IPD: No